CLINICAL TRIAL: NCT02705274
Title: Panretinal Photocoagulation Versus Intravitreal Bevacizumab for Proliferative Diabetic Retinopathy
Brief Title: PRP vs Bevacizumab for PDR Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Marashi Eye Clinic (Other)
Responsible Party: Principal Investigator, Ameen Marashi, MD, Ophthalmologist Retina specialist, Marashi Eye Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol PDR 1
Record Dates: First submitted 2016-02-29; First posted 2016-03-10 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Bevacizumab

ARMS (2):
- Prompt Panretinal Photocoagulation (Active Comparator): PRP= Panretinal Photocoagulation. PRP alone.
  Interventions: Procedure: Panretinal photocoagulation
- Bevacizumab with deferred PRP (Experimental): Bevacizumab = Anti vascular endothelial growth factor. PRP= Panretinal photocoagulation. Intravitreal anti-VEGF with PRP only if indicated.
  Interventions: Drug: Bevacizumab; Procedure: Panretinal photocoagulation

INTERVENTIONS:
Drug: Bevacizumab — Drug: 1.25-mg Bevacizumab Intravitreal injection of 1.25 mg Bevacizumab at baseline and up to every 4 weeks using defined retreatment criteria.
  Other: Deferred panretinal photocoagulation PRP is deferred until failure/futility criteria for intravitreal injection are met.
  Arms: Bevacizumab with deferred PRP
Procedure: Panretinal photocoagulation — Panretinal photocoagulation (full session completed within 42 days).

SUMMARY:
Protocol S by DRCR.net has shown that receive Ranibizumab as anti-vascular endothelial growth factor (anti-VEGF) therapy with deferred panretinal photocoagulation (PRP) are non-inferior to those in eyes that receive standard prompt PRP therapy, however with some visual functional benefits and less complications with Ranibizumab arm.

Applying Protocol S in real world scenario may add cost burden to the patient as patients need about 7 injections per year which will cost the patient about 7000 US dollars a year as minimum The primary objective of this protocol is to determine the visual acuity outcomes at 1 year in eyes with proliferative diabetic retinopathy (PDR) using Bevacizumab 1.25 mg instead of Ranbizumab to lower the cost burden

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Presence of PDR which the investigator intends to manage with PRP alone but for which PRP can be deferred for at least 4 weeks in the setting of intravitreal Bevacizumab , in the investigator's judgment.
* Best corrected Snellen equivalent 20/320 or higher on the day of randomization.
* Media clarity, pupillary dilation, and study participant cooperation sufficient to administer PRP and obtain adequate fundus photographs and OCT.

Exclusion Criteria:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization
* Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years.
* Tractional retinal detachment involving the macula. -- A tractional retinal detachment is not an exclusion if it is outside of the posterior pole (not threatening the macula) and in the investigator's judgment, is not a contraindication to intravitreal Bevacizumab treatment and also does not preclude deferring PRP for at least 4 weeks in the setting of intravitreal Bevacizumab
* Macular edema is present that is considered to be related to ocular surgery such as cataract extraction orclinical exam and/or OCT suggest that vitreoretinal interface abnormalities disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of any macular edema.
* An ocular condition is present (other than diabetic retinopathy) that, in the opinion of the investigator, might alter visual acuity during the course of the study (e.g., retinal vein or artery occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma,
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye were otherwise normal).
* History of intravitreal anti-VEGF treatment at any time in the past 2 months.
* History of corticosteroid treatment (intravitreal ) at any time in the past 4 months.
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
* Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis
* Uncontrolled glaucoma (in investigator's judgment).
* Aphakia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Proportion of visual acuity improvement using Snellen chart or equivalent from baseline and 1 year | 1 year

SECONDARY OUTCOMES:
Amount of treatment cost | 1 year
Percent of eyes with vitreous hemorrhage | 1 year
Proportion of eyes with complete regression of neovascularization on fundus photograph | 1 year
Proportion of eyes with progression to central subfield involved diabetic macular edema | 1 year
Proportion of eyes Need for Vitrectomy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ameen Marashi, MD, Principal Investigator — Marashi Eye Clinic
Locations (1):
- Marashi Eye Clinic, Aleppo, Syria

REFERENCES:
- [Result] Marashi A, Abukhalaf I, Alfaraji R, Choman Y, Salahieh A (2017) Panretinal Photocoagulation versus Intravitreal Bevacizumab for Proliferative Diabetic Retinopathy Treatment. Adv Ophthalmol Vis Syst 7(1): 00211. DOI: 10.15406/aovs.2017.07.00211
- See also: Marashi A, Abukhalaf I, Alfaraji R, Choman Y, Salahieh A (2017) Panretinal Photocoagulation versus Intravitreal Bevacizumab for Proliferative Diabetic Retinopathy Treatment. Adv Ophthalmol Vis Syst 7(1): 00211. DOI: 10.15406/aovs.2017.07.00211 — http://medcraveonline.com/AOVS/AOVS-07-00211.pdf